CLINICAL TRIAL: NCT00000559
Title: Women's Estrogen/Progestin Lipid Lowering Hormone Atherosclerosis Regression Trial (WELL-HART)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 103
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2005-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Estrogen Replacement Therapy; Hormone Replacement Therapy; Estradiol; Medroxyprogesterone

INTERVENTIONS:
Drug: estrogen replacement therapy
Drug: hormone replacement therapy
Drug: estradiol
Drug: medroxyprogesterone

SUMMARY:
To determine the effects, in postmenopausal women, of hormone replacement therapy on progression/regression of coronary heart disease, as measured by quantitative angiography.

DETAILED DESCRIPTION:
BACKGROUND:

The trial was a logical extension of preceding observational and cross-sectional studies on estrogen replacement therapy. Overall, the studies suggested a 50 percent reduction in risk of coronary heart disease in current estrogen users compared to non-users. In spite of such striking findings, most studies had been prone to a number of biases. One major criticism of observational studies had been that women receiving estrogen were generally healthier and more compliant than non-estrogen users.

There was a very large body of observational data suggesting that the use of estrogen in postmenopausal women reduced coronary heart disease mortality by approximately 45 percent. At the same time, there had been some concern that replacement therapy increased the likelihood of uterine cancer and perhaps breast cancer as well, although it was generally accepted that this risk was probably significantly less than the benefits obtained from the reduction of coronary heart disease mortality.

DESIGN NARRATIVE:

Randomized, double-blind, placebo-controlled. After baseline angiograms, patients were randomized to one of three arms: micronized 17-beta estradiol, 1 milligram per day; 17-beta estradiol plus medroxyprogesterone, 5 milligrams per day for twelve days per month; and placebo. Subjects in all three arms received lipid-lowering therapy, low fat/low cholesterol diet, and the HMG-CoA reductase inhibitor, pravastatin, in sufficient dosage to reduce low density lipoprotein (LDL) cholesterol levels below 130 mg/dl. The primary endpoint was progression/regression of coronary obstructive disease as measured by angiography, including the expert human panel and quantitative computer analysis. The secondary endpoint was carotid media-intima thickness determined by ultrasound. Clinical measures included lipids, lipoproteins, apolipoproteins, estradiol and medroxyprogesterone levels, urinary prostanoid metabolites, and insulin/glucose metabolism. Subjects were recruited at three centers with active coronary angiography units. Several core facilities supported the study: a Core Lipid Lab, a Reproductive Endocrine Lab, the Biostatistics Lab (Data Coordinating Center) and the Angiographic Imaging Laboratory.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Postmenopausal women with angiographically-documented coronary disease. Approximately 70 percent minority

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-03; Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hodis — University of Southern California

REFERENCES:
- [Background] Slater CC, Zhang C, Hodis HN, Mack WJ, Boostanfar R, Shoupe D, Paulson RJ, Stanczyk FZ. Comparison of estrogen and androgen levels after oral estrogen replacement therapy. J Reprod Med. 2001 Dec;46(12):1052-6. PMID 11789085
- [Background] Wilcox JG, Hwang J, Hodis HN, Sevanian A, Stanczyk FZ, Lobo RA. Cardioprotective effects of individual conjugated equine estrogens through their possible modulation of insulin resistance and oxidation of low-density lipoprotein. Fertil Steril. 1997 Jan;67(1):57-62. doi: 10.1016/s0015-0282(97)81856-0. PMID 8986684
- [Background] Hodis HN, Mack WJ, Azen SP, Lobo RA, Shoupe D, Mahrer PR, Faxon DP, Cashin-Hemphill L, Sanmarco ME, French WJ, Shook TL, Gaarder TD, Mehra AO, Rabbani R, Sevanian A, Shil AB, Torres M, Vogelbach KH, Selzer RH; Women's Estrogen-Progestin Lipid-Lowering Hormone Atherosclerosis Regression Trial Research Group. Hormone therapy and the progression of coronary-artery atherosclerosis in postmenopausal women. N Engl J Med. 2003 Aug 7;349(6):535-45. doi: 10.1056/NEJMoa030830. PMID 12904518
- [Derived] Steiner AZ, Xiang M, Mack WJ, Shoupe D, Felix JC, Lobo RA, Hodis HN. Unopposed estradiol therapy in postmenopausal women: results from two randomized trials. Obstet Gynecol. 2007 Mar;109(3):581-7. doi: 10.1097/01.AOG.0000251518.56369.eb. PMID 17329508